CLINICAL TRIAL: NCT01738763
Title: Effects of Different Doses of Pinitol on Carbohydrate Metabolism Parameters in Healthy Subjects: a Randomized Cross-over Placebo-controlled Study
Brief Title: Effects of Different Doses of Pinitol on Carbohydrate Metabolism Parameters in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Antonio Hernández Mijares, PhD, MD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: WIL-PIN-2011-01
Record Dates: First submitted 2012-11-20; First posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Healthy; Insulin Sensitivity
Keywords: Glucose; Insulin; 3-O-methyl-D-chiro-inositol
MeSH Terms: conditions — Insulin Resistance | interventions — pinitol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low dose (2.5 g of pinitol) (Experimental): Each subject completed two 1-day trials separated by a 1-week interval. The subjects were randomized by alternation method to belong to the group of low, intermediate or high dose, containing 2.5, 4.0 or 6.0 g of pinitol, respectively. Each subject was newly randomized (1:1) and cross-over into one of two groups: one that received the pinitol-enriched beverage, and the other a placebo beverage. In this way, each dose and its corresponding placebo were studied in 10 normoglycaemic subjects.
  Interventions: Dietary Supplement: Pinitol
- Intermediate dose (4.0 g of pinitol) (Experimental): Each subject completed two 1-day trials separated by a 1-week interval. The subjects were randomized by alternation method to belong to the group of low, intermediate or high dose, containing 2.5, 4.0 or 6.0 g of pinitol, respectively. Each subject was newly randomized (1:1) and cross-over into one of two groups: one that received the pinitol-enriched beverage, and the other a placebo beverage. In this way, each dose and its corresponding placebo were studied in 10 normoglycaemic subjects.
  Interventions: Dietary Supplement: Pinitol
- High dose (6.0 g of pinitol) (Experimental): Each subject completed two 1-day trials separated by a 1-week interval. The subjects were randomized by alternation method to belong to the group of low, intermediate or high dose, containing 2.5, 4.0 or 6.0 g of pinitol, respectively. Each subject was newly randomized (1:1) and cross-over into one of two groups: one that received the pinitol-enriched beverage, and the other a placebo beverage. In this way, each dose and its corresponding placebo were studied in 10 normoglycaemic subjects.
  Interventions: Dietary Supplement: Pinitol

INTERVENTIONS:
Dietary Supplement: Pinitol — Three doses of Fruit Up® (diluted with mineral water to a final volume of 330 ml) were evaluated, and were equivalent to an intake of 2.5, 4.0 and 6.0 g of pinitol. The placebo beverage contained equal amounts of non-polyol carbohydrates with similar macronutrient composition and energy intake as that those obtained through the pinitol beverage, but excluding pinitol.
  Other Names: 3-O-methyl-D-chiro-inositol

SUMMARY:
The purpose of this study was to assess the acute effects of increasing doses of pinitol on glucose tolerance and insulin sensitivity and to evaluate the absorption of pinitol after consumption of an oral nutritive pinitol-enriched beverage in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for all subjects were age range of 18-65 years, body mass index of 20-30 Kg/m2 and clinically normal kidney function, liver function, heart function, protein status and haematological profile.

Exclusion Criteria:

* Exclusion criteria were pregnancy or lactation, alteration of carbohydrate metabolism, fasting glycaemia ≥5.55 mmol/l on at least two previous occasions, diabetes, or medication known to interfere with glucose metabolism.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Dose-response curves to assess the change in glucose and insulin concentration after an oral ingestion of different doses of pinitol with respect to the corresponding placebo | up to 120 minutes
  Each subject attended the Endocrinology Service in the morning after 12-hour overnight fasting. Blood sample was collected in vacutainer serum separator tubes at baseline (minute 0; while still fasting), 15, 30, 45, 60, 90 and 120 minutes after consumption of the tested product placebo or pinitol-enriched beverage. Glucose concentrations were measured by means of enzymatic assay in an autoanalyzer. Insulin concentrations were determined by enzyme-linked immunosorbent assay.

SECONDARY OUTCOMES:
Dose-response curves to assess the change in pinitol concentration after an oral ingestion of different doses of pinitol with respect to the corresponding placebo | up to 240 minutes
  Plasma pinitol analysis blood samples were collected into vacutainers containing lithium heparin at baseline, 60, 120, 180 and 240 minutes after consumption of the tested product placebo or pinitol-enriched beverage. Pinitol concentration was determined by gas chromatography/ mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Hernández Mijares, MD, PhD, Principal Investigator — University of Valencia
Locations (1):
- University Hospital Dr Peset, Valencia, Spain

REFERENCES:
- [Background] Stull AJ, Wood KV, Thyfault JP, Campbell WW. Effects of acute pinitol supplementation on plasma pinitol concentration, whole body glucose tolerance, and activation of the skeletal muscle insulin receptor in older humans. Horm Metab Res. 2009 May;41(5):381-6. doi: 10.1055/s-0028-1128140. Epub 2009 Feb 16. PMID 19221977
- [Background] Campbell WW, Haub MD, Fluckey JD, Ostlund RE Jr, Thyfault JP, Morse-Carrithers H, Hulver MW, Birge ZK. Pinitol supplementation does not affect insulin-mediated glucose metabolism and muscle insulin receptor content and phosphorylation in older humans. J Nutr. 2004 Nov;134(11):2998-3003. doi: 10.1093/jn/134.11.2998. PMID 15514265
- [Background] Larner J, Allan G, Kessler C, Reamer P, Gunn R, Huang LC. Phosphoinositol glycan derived mediators and insulin resistance. Prospects for diagnosis and therapy. J Basic Clin Physiol Pharmacol. 1998;9(2-4):127-37. doi: 10.1515/jbcpp.1998.9.2-4.127. PMID 10212830
- [Background] Larner J, Brautigan DL, Thorner MO. D-chiro-inositol glycans in insulin signaling and insulin resistance. Mol Med. 2010 Nov-Dec;16(11-12):543-52. doi: 10.2119/molmed.2010.00107. Epub 2010 Aug 27. PMID 20811656
- [Background] Kang MJ, Kim JI, Yoon SY, Kim JC, Cha IJ. Pinitol from soybeans reduces postprandial blood glucose in patients with type 2 diabetes mellitus. J Med Food. 2006 Summer;9(2):182-6. doi: 10.1089/jmf.2006.9.182. PMID 16822203
- [Background] Kim JI, Kim JC, Kang MJ, Lee MS, Kim JJ, Cha IJ. Effects of pinitol isolated from soybeans on glycaemic control and cardiovascular risk factors in Korean patients with type II diabetes mellitus: a randomized controlled study. Eur J Clin Nutr. 2005 Mar;59(3):456-8. doi: 10.1038/sj.ejcn.1602081. PMID 15536472
- [Background] Kim HJ, Park KS, Lee SK, Min KW, Han KA, Kim YK, Ku BJ. Effects of pinitol on glycemic control, insulin resistance and adipocytokine levels in patients with type 2 diabetes mellitus. Ann Nutr Metab. 2012;60(1):1-5. doi: 10.1159/000334834. Epub 2011 Dec 16. PMID 22179130